CLINICAL TRIAL: NCT01864915
Title: Prucalopride + Prucalopride Booster vs. Prucalopride + Picosalax Booster for the Colon Capsule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Hotel Dieu Hospital (Other); Janssen Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Lawrence Hookey, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: DMED 1578-13 HOOKEY; 9427-D2773-21C (Other: Health Canada TPD)
Record Dates: First submitted 2013-05-25; First posted 2013-05-30 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Bowel Cleansing; Colon Capsule Completion Times
Keywords: colon capsule; bowel preparation; booster; prucalopride; picosalax
MeSH Terms: interventions — prucalopride

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No Booster-low dose prucalopride booster (Experimental): low dose prucalopride booster arm
  Interventions: Drug: Prucalopride; Procedure: Colon Capsule
- Prucalopride Booster-high dose prucalopride booster (Experimental): additional 2mg prucalopride at time of capsule ingestion
  Interventions: Drug: Prucalopride; Procedure: Colon Capsule
- Picosalax Booster Arm (Experimental): One sachet of Picosalax 2hrs after capsule ingestion and 1/2 sachet at 4 hrs after swallowing colon capsule.
  Interventions: Drug: Prucalopride; Procedure: Colon Capsule

INTERVENTIONS:
Drug: Prucalopride — Prucalopride 2mg daily starting three days before the colon capsule study (total of 4 doses with the last at 0800hrs on day of colon capsule study)
  Other Names: RESTORAN
Procedure: Colon Capsule — Colon capsule procedure performed day prior to colonoscopy, at 0800 hrs on day 4.

SUMMARY:
Colon capsule endoscopy is a new technology that is a noninvasive method of examining the large bowel. The bowel preparation required for this test differs from colonoscopy in that it needs to clean the colon but also needs to provide propulsion. Most published studies have used medications as part of their regime that are not available in parts of North America (ex. sodium phosphate) and have shown poor test completion, bowel preparation and polyp detection rates.

Objective: In this study a bowel preparation for the colon capsule is proposed that uses medications approved for use in Canada that may provide a better preparation quality and better completion rates.

Methods: Patients who are being referred for a colonoscopy will be recruited to participate in the study. They will all receive split-dose polyethylene glycol (PEG) for bowel preparation. They will be randomized to receive either 1) Prucalopride 2mg daily for four days, 2) Prucalopride 2mg daily for four days plus a Prucalopride booster, or 3) Prucalopride 2mg for four days plus 1 and 1/2 sachets of Picosalax boosters for the colon capsule study. The day after the colon capsule they will drink PEG ( 2 Liters) at 5am -or approx 4hrs prior to procedure time and return for a colonoscopy. The colon capsule results will be reviewed by two endoscopists experienced in video capsule endoscopy who will assess the bowel preparation using a previously defined scale and examine for polyps. We propose that administering Prucalopride daily for 4 days will increase intestinal motility and improve colon capsule completion rates and a booster dose of Picosalax will improve colon capsule completion rates compared to prucalopride by itself.

DETAILED DESCRIPTION:
Colon capsule endoscopy is a new technology that is a noninvasive method of examining the large bowel. The bowel preparation required for this test differs from colonoscopy in that it needs to clean the colon but also needs to provide propulsion. Most published studies have used medications as part of their regime that are not available in parts of North America (ex. sodium phosphate) and have shown poor test completion, bowel preparation and polyp detection rates.

Objective: In this study a bowel preparation for the colon capsule is proposed that uses medications approved for use in Canada that may provide a better preparation quality and better completion rates.

Methods: Patients who are being referred for a colonoscopy will be recruited to participate in the study. They will all receive split-dose polyethylene glycol (PEG) for bowel preparation. They will be randomized to receive either 1) Prucalopride 2mg daily for four days, 2) Prucalopride 2mg daily for four days plus a Prucalopride booster, or 3) Prucalopride 2mg for four days plus 1 and 1/2 sachets of Picosalax boosters for the colon capsule study. The day after the colon capsule they will drink PEG ( 2 Liters) at 5am -or approx 4hrs prior to procedure time and return for a colonoscopy. The colon capsule results will be reviewed by two endoscopists experienced in video capsule endoscopy who will assess the bowel preparation using a previously defined scale and examine for polyps. We propose that administering Prucalopride daily for 4 days will increase intestinal motility and improve colon capsule completion rates and a booster dose of Picosalax will improve colon capsule completion rates compared to prucalopride by itself

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-75 being referred for colonoscopy

Exclusion Criteria:

* symptoms of dysphagia or any problems with swallowing, bowel obstruction or ileus, known stricture or fistula, inflammatory bowel disease, previous small or large bowel surgery, severe gastroparesis or motility disorder, severe renal impairment ( defined as lab test result eGFR ie. estimated Glomerular Filtration Rate less than 55 within three months of study), congestive heart failure (NYHA III or IV), ischemic heart disease (acute event in the last 6mths), decompensated cirrhosis or severe hepatic dysfunction (ascites or known lab test INR>2), history of serious arrhythmia or any other severe and clinically unstable concomitant disease (eg. lung disease, neurological or psychiatric disorder, cancer, AIDS and other endocrine disorder) ,diabetics on treatment with insulin or hypoglycemic, pregnant or nursing women, galactose intolerance (since the tablets contain lactose monohydrate, patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose/galactose malabsorption must not take this medicinal product.) or known hypersensitivity to the drug or to any ingredient in the formulation (each 2mg tablet contains prucalopride 2 mg. Nonmedicinal ingredients: tablet core: lactose monohydrate, microcrystalline cellulose, colloidal silicon dioxide, and magnesium stearate; coating: hypromellose, lactose monohydrate, triacetin, titanium dioxide, macrogol 3000, iron oxide red, iron oxide yellow, and FD&C Blue No. 2 Aluminum Lake) Females of child bearing potential who are unwilling to use appropriate birth control methods during the study will not be able to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To assess the quality of the bowel preparations | Day of colon capsule procedure and day of colonoscopy
  Colon capsule bowel prep assessed with previously used scale completed by designated gastroenterologists.
  Colonoscopy bowel prep assessed by completion of Aronchick Scale by endoscopist performing procedure.

SECONDARY OUTCOMES:
Tolerance of Bowel Preparation with survey | Day of colonoscopy
Gastric, small bowel and colon transit time | Day of colon capsule

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hookey, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
final analysis dataset shared with Janssen Inc (study sponsor)